CLINICAL TRIAL: NCT00271505
Title: A Phase II Evaluation of Avastin in Combination With Docetaxel and Carboplatin as Chemotherapy in Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: Avastin/Docetaxel/Carboplatin in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0224; NCI-2012-01621 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; Bevacizumab; Carboplatin; Docetaxel; Avastin; NSCLC; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Paraplatin®; Taxotere
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avastin + Docetaxel + Carboplatin (Experimental): Avastin 15 mg/kg intravenously (IV) every 3 weeks. Docetaxel 75 mg/m2 IV every 3 weeks. Carboplatin AUC 6 IV every 3 weeks.
  Interventions: Drug: Bevacizumab (Avastin); Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — 15 mg/kg intravenously (IV) every 3 weeks
  Other Names: Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Carboplatin — AUC 6 IV every 3 weeks
  Other Names: Paraplatin®
Drug: Docetaxel — 75 mg/m2 IV every 3 weeks
  Other Names: Taxotere

SUMMARY:
The goal of this clinical research study is to evaluate the effectiveness of Avastin® in combination with docetaxel and carboplatin in the treatment of lung cancer. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Avastin® is a humanized monoclonal antibody that binds to vascular endothelial growth factor (VEGF). VEGF plays an important role in the growth of both normal and abnormal blood vessels. Avastin® is designed to prevent or slow down the growth of cancer cells by blocking the effects of VEGF.

Docetaxel and carboplatin are standard chemotherapy drugs that have been approved by the FDA for the treatment of NSCLC. Docetaxel and carboplatin are designed to work by stopping the division of cancer cells.

If you are found to be eligible, you will begin receiving Avastin®, docetaxel, and carboplatin. Avastin®, carboplatin, and docetaxel will be given by vein once every 3 weeks. The first dose of Avastin® will be given over 90 minutes. The second dose of Avastin® will be given over 60 minutes. All other doses of Avastin® will be given over 30 minutes. Carboplatin and docetaxel will always be given over 30 minutes. They will be given on the same day every 3 weeks (1 cycle). You may receive up to 6 cycles of treatment. You will receive standard premedication with dexamethasone to help decrease the risk of side effects. Dexamethasone will be taken before you receive your docetaxel infusion.

During the study, you will have blood tests (about 2 teaspoons) every 3 weeks to look at your blood counts. These samples will be used only for routine lab tests. You will be seen by a physician every 3 weeks and given a physical exam. Your blood pressure will be monitored, and you will be asked about any side effects you are experiencing. A performance status evaluation will also be done. In addition, you will have a urine test every 2 cycles of treatment.

After 2 cycles of treatment (6 weeks), you will have a chest x-ray and computerized tomography (CT) or magnetic resonance imaging (MRI) scan to evaluate the status of the disease. These will be repeated every 2 cycles. Your continued participation in this study depends on how your cancer responds to the study drugs. Your doctor may decide to take you off this study if you experience significant side effects or your medical condition worsens. You may continue receiving bevacizumab for as long as your cancer responds to study treatment.

You will be followed-up on by phone or at routine clinic visits for at least 12 months to monitor your condition and disease status.

This is an investigational study. Avastin® has been approved by the FDA for the treatment of colorectal cancer. Docetaxel and carboplatin are FDA approved and commercially available. The use of these drugs together in this study is experimental. A total of 50 patients will take part in this study. All participants will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, at least 18 years old, with histologically confirmed, advanced stage IIIB or IV NSCLC for whom no curative options exist and for whom docetaxel and carboplatin is a reasonable treatment option;
2. At least 1 target lesion that is unidimensionally measurable as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) and has not been previously irradiated;
3. Eastern Cooperative Oncology Group Performance Status of 0 or 1, (determined within 2 weeks prior to receiving study medication;
4. Ability to understand and adhere to the protocol requirements, and give informed consent
5. Use of effective means of contraception (men and women) in subjects of child-bearing potential. Child-bearing potential is defined as follows: A woman of childbearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Patients who have had docetaxel in nonradiosensitizing therapy
2. Patients who have received prior full dose systemic chemotherapy for NSCLC (ie neoadjuvant, adjuvant, or metastatic) within the last 6 months.
3. Eastern Cooperative Oncology Group (ECOG) status of 2 or greater
4. Screening clinical laboratory values:*absolute neutrophil count (ANC) of <1,500/µL *Platelet count of <75,000/µL * international normalized ratio (INR) >/= 1.5 *T bilirubin elevation above normal (MDACC upper normal limit is 1.0 mg/dL) *Serum creatinine of >2.0 mg/dL *Hemoglobin of <9 mg/dL (may be transfused or receive epoetin alfa [e.g., Epogen®] to maintain or exceed this level) *The pt is ineligible if: 1.alk phos>5xULN; 2.AST or ALT >5xULN; 3.alk phos >1xULN but </= 2.5xULN AND AST or ALT >1.5xULN but </=5xULN;4.alk phos >2.5xULN but </=5xULN AND AST or ALT > 1xULN but</= 1.5xULN; 5.alk phos >2.5xULN but</=5xULN AND AST or ALT >1.5xULN but </=5xULN
5. Inability to comply with study and/or follow-up procedures
6. History of other disease, active infection, metabolic dysfunction , physical examination finding, or clinical laboratory finding which is uncontrolled requiring medical intervention giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
7. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a bevacizumab cancer study
8. Prior exposure to anti-VEGF therapy
9. Blood pressure of > 140/90 mmHg as documented in two consecutive blood pressure readings within 4 hours
10. Any prior history of hypertensive crisis or hypertensive encephalopathy
11. New York Heart Association (NYHA) Grade II or greater congestive heart failure
12. History of myocardial infarction or unstable angina within 6 months
13. History of stroke or transient ischemic attack within 6 months
14. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
15. Evidence of bleeding diathesis or coagulopathy
16. Presence of central nervous system or brain metastases at any time
17. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
18. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
19. Pregnant (positive pregnancy test) or lactating
20. Proteinuria at screening as demonstrated by either: Urine protein:creatinine (UPC) ratio > 1.0 at screening OR Urine dipstick for proteinuria > 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < 1g of protein in 24 hours to be eligible).
21. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
22. Serious, non-healing wound, ulcer, or bone fracture
23. Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, cavitation.
24. History of hemoptysis (bright red blood of 1/2 teaspoon or more)
25. Full dose anticoagulation, chronic use of Aspirin (>325 mg/day) or NSAIDs
26. Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-12-05 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vali Papadimitrakopoulou, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was interrupted before the planned 50 patients were enrolled because of slow accrual after bevacizumab became commercially available in the United States for NSCLC treatment.
Groups:
- Carboplatin (AUC 6), Docetaxel (75 mg/m2), and Bevacizumab (: Patients were treated with up to 6 cycles of carboplatin (AUC 6), docetaxel (75 mg/m2), and bevacizumab (15 mg/kg) on Day 1 every 21 days. Patients with an objective response or stable disease received maintenance bevacizumab (15 mg/kg) every 21 days until disease progression. The primary endpoint was median progression-free survival. Six cycles of chemotherapy plus bevacizumab were planned. Patients who demonstrated stable disease (SD), partial response (PR), or complete response (CR) to treatment continued on single-agent bevacizumab 15 mg/kg every 21 days until disease progression or intolerable toxicity. Patients who discontinued chemotherapy before 6 cycles of treatment were also allowed to continue on single-agent bevacizumab in the absence of progressive disease (PD).
Period: Overall Study
Arm/Group | Carboplatin (AUC 6), Docetaxel (75 mg/m2), and Bevacizumab (
Started | 43
Completed | 38
Not Completed | 5
Not completed — Screen Failure | 3
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population differs from the number of participants in that the BAP does not account for the 3 patients who signed consent and screened out of the study.
Groups:
- Carboplatin, Docetaxel, and Bevacizumab: Forty patients were treated with up to 6 cycles of carboplatin (AUC 6), docetaxel (75 mg/m2), and bevacizumab (15 mg/kg) on Day 1 every 21 days. Patients with an objective response or stable disease received maintenance bevacizumab (15 mg/kg) every 21 days until disease progression. The primary endpoint was median progression-free survival. Six cycles of chemotherapy plus bevacizumab were planned. Patients who demonstrated stable disease (SD), partial response (PR), or complete response (CR) to treatment continued on single-agent bevacizumab 15 mg/kg every 21 days until disease progression or intolerable toxicity. Patients who discontinued chemotherapy before 6 cycles of treatment were also allowed to continue on single-agent bevacizumab in the absence of progressive disease (PD).
Arm/Group | Carboplatin, Docetaxel, and Bevacizumab
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression-Free Survival (PFS)
Description: Bevacizumab has recently been demonstrated to prolong overall survival when added to carboplatin and paclitaxel for chemotherapy-naı¨ve patients with nonsquamous nonsmall-cell lung cancer (NSCLC). However, the effects of combining bevacizumab with other standards, front-line, platinum-based doublets have not been extensively explored.We designed this single treatment arm, phase 2 trial to determine whether the combination of carboplatin, docetaxel, and bevacizumab is tolerable and prolongs progression-free survival of chemotherapy-naı¨ve patients with advanced, on squamous NSCLC.
Time Frame: Baseline up to 12 months or disease progression/death
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carboplatin, Docetaxel, and Bevacizumab: Up to 6 cycles of carboplatin (AUC 6), Tocetaxel (75 mg/m2), and Bevacizumab (15 mg/kg) on Day 1 every 21 days
Arm/Group | Carboplatin, Docetaxel, and Bevacizumab
Number analyzed (Participants) | 38
months | 7.9 [6.0 to 11.1]

2. Secondary Outcome: Overall Survival (OS)- 5 Years
Description: Secondary endpoints of the study included the assessment of overall survival, disease control rate (CR þPR þ SD, defined by RECIST16), and evaluation of the safety profile of this triple-agent regimen. All patients who received at least 1 dose of the study drug were analyzed for efficacy and toxicity endpoints.
Time Frame: Baseline start of treatment to death, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carboplatin,Docetaxel, and Bevacizumab: Up to 6 cycles of carboplatin (AUC 6), Tocetaxel (75 mg/m2), and Bevacizumab (15 mg/kg) on Day 1 every 21 days"
Arm/Group | Carboplatin,Docetaxel, and Bevacizumab
Number analyzed (Participants) | 40
months | 16.5 [13.6 to 31.2]

3. Secondary Outcome: Disease Control Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1 .0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)= CR+ PR.
Time Frame: Baseline start of treatment to death, assessed up to 6 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carboplatin,Docetaxel, and Bevacizumab
Number analyzed (Participants) | 40
percentage of participants | 95 [88 to 100]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Groups:
- Carboplatin,Docetaxel, and Bevacizumab: Up to 6 cycles of carboplatin (AUC 6), Tocetaxel (75 mg/m2), and Bevacizumab (15 mg/kg) on Day 1 every 21 days
Arm/Group | Carboplatin,Docetaxel, and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 13/40
Other Adverse Events (participants affected / at risk) | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin,Docetaxel, and Bevacizumab (N=40)
Hemoptysis (Blood and lymphatic system disorders) | 1
Pulmonary Hemmorhage (Respiratory, thoracic and mediastinal disorders) | 1
embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (Blood and lymphatic system disorders) | 1
Perforation Duodenum G4 (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Rt Ing Hernia (Gastrointestinal disorders) | 1
Fatigue & Infection G3 (Blood and lymphatic system disorders) | 1
Mild Anemia of Chronic Disease and Fatigue (Blood and lymphatic system disorders) | 1
Sudden Death (General disorders) | 1
Death (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin,Docetaxel, and Bevacizumab (N=40)
Anemia (Blood and lymphatic system disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 25
Anorexia (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 21
Nail Change (Skin and subcutaneous tissue disorders) | 13
Hyperglycemia (Endocrine disorders) | 21
Hypomagnesemia (Metabolism and nutrition disorders) | 20
Nausea (Gastrointestinal disorders) | 15
Stomatitis (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT00271505/Prot_SAP_000.pdf